CLINICAL TRIAL: NCT05364762
Title: Single Center Pilot Study to Investigate the Efficacy of Adding Itacitinib to Post-Transplant Cyclophosphamide as Graft-Versus-Host Disease Prophylaxis After Reduced Intensity Conditioning Matched Donor Hematopoietic Cell Transplantation With Peripheral Blood Stem Cells as Graft Source
Brief Title: Adding Itacitinib to Cyclophosphamide and Tacrolimus for the Prevention of Graft Versus Host Disease in Patients Undergoing Hematopoietic Stem Cell Transplants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21776; NCI-2022-03765 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21776 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Myeloproliferative Disorders; Primary Myelofibrosis | interventions — Cyclophosphamide; itacitinib; INCB039110; Peripheral Blood Stem Cell Transplantation; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (PBSCs, cyclophosphamide, itacitinib, tacrolimus) (Experimental): Patients undergo peripheral blood stem cell infusion on day 0. Patients receive cyclophosphamide IV QD on days 3 and 4, itacitinib PO QD on days 5-100, and tacrolimus IV or PO on days 6-65.
  Interventions: Drug: Cyclophosphamide; Drug: Itacitinib; Procedure: Peripheral Blood Stem Cell Transplantation; Other: Quality-of-Life Assessment; Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Itacitinib — Given PO
  Other Names: INCB 039110; INCB-039110; INCB039110
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood stem cell infusion
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This clinical trial evaluates the safety and effectiveness of adding itacitinib to cyclophosphamide and tacrolimus for the prevention of graft versus host disease (GVHD) in patients undergoing hematopoietic stem cell transplant. Itacitinib is an enzyme inhibitor that may regulate the development, proliferation, and activation of immune cells important for GVHD development. Cyclophosphamide and tacrolimus are immunosuppressive agents that may prevent GVHD in patients who receive stem cell transplants. Giving itacitinib in addition to cyclophosphamide and tacrolimus may be more effective at preventing GVHD in patients receiving hematopoietic stem cell transplants.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Safety lead-in: Determine if shortening tacrolimus administration period to 60 days (day +65 post-hematopoietic cell transplantation [HCT]), when combined with post-transplant cyclophosphamide (PTCy) and itacitinib at a fixed dose level as graft-versus-host disease (GVHD) prophylaxis, is safe and effective after mobilized peripheral blood stem cell (PBSC) allogeneic hematopoietic cell transplantation (HCT) from a matched related/unrelated donor, as assessed by grade 3-4 GVHD as dose limiting toxicity.

II. Following the safety lead-in, evaluate the efficacy of PTCy, itacitinib and tacrolimus GVHD prophylaxis, as assessed by 1-year GVHD-free relapse-free survival (GRFS).

SECONDARY OBJECTIVES:

I. Evaluate the safety of this regimen by assessing:

Ia. Adverse events: type, frequency, severity, attribution, time course, duration.

Ib. Complications including acute and chronic GVHD, infections and delayed engraftment.

II. Estimate overall survival (OS), progression-free survival (PFS), cumulative incidences of relapse/disease progression, and non-relapse mortality (NRM) at 100 days, and 1-year post-transplant.

III. Estimate rates of acute and chronic GvHD, infections, and neutrophil recovery.

EXPLORATORY OBJECTIVES:

I. Donor cell engraftment will be assessed by count monitoring and short tandem repeat (STR) chimerism analysis on days +30 and day +100.

II. Describe the kinetics of immune cell recovery. III. Evaluate patient's quality of life on day +100, 6 months and one-year post-HCT.

IV. Pharmacokinetics: serial blood sampling will be done to evaluate the steady-state pharmacokinetics of itacitinib after PTCy.

V. Describe the kinetics of GVHD biomarkers, JAK-related inflammatory cytokines and STAT phosphorylation.

VI. Evaluate and describe the cytokine release syndrome (CRS) post-HCT by assessing the incidence, frequency, and severity of CRS.

VII. Obtain a preliminary estimate of gut microbiome diversity at baseline (preferably before fludarabine administration), and then on days +14, +30, and +100.

OUTLINE:

Patients undergo peripheral blood stem cell infusion on day 0. Patients receive cyclophosphamide intravenously (IV) once daily (QD) on days 3 and 4, itacitinib orally (PO) QD on days 5-100, and tacrolimus IV or PO on days 6-65.

After completion of study treatment, patients are followed up at day 180 and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: =< 80 years

  * Note: Patients > 70 years of age must have Karnofsky performance status >= 80 and HCT-comorbidity index (CI) =< 2
* Karnofsky performance status >= 70%
* Patients with the following diagnosis, eligible to undergo allogeneic HCT from an 8/8 match related/unrelated donor (A, B, C, DR by high resolution typing)

  * Acute leukemias (acute myeloid leukemia [AML] or acute lymphoblastic leukemia [ALL]) in complete remission with bone marrow (BM) blast of < 5%
  * Myelofibrosis (MF): Primary or secondary with high- or intermediate-2 risk per Dynamic International Prognostic Scoring System (DIPSS)
  * Myelodysplastic syndrome (blast < 10%)
  * Myeloproliferative neoplasm (MPN) other than MF needing HCT
  * Chronic myelomonocytic leukemia (CMML)
* Total bilirubin =< 2 x upper limit of normal (ULN) (unless has Gilbert's disease) (within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 5 x ULN (within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Creatinine clearance of >= 60 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 30 days prior to day 1 of protocol therapy unless otherwise stated)
* Left ventricular ejection fraction (LVEF) >= 50%

  * Note: To be performed within 30 days prior to day 1 of protocol therapy
* If able to perform pulmonary function tests: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC) and diffusion capacity of the lungs for carbon monoxide (DLCO) (diffusion capacity) >= 50% of predicted (corrected for hemoglobin) (within 30 days prior to day 1 of protocol therapy)
* If unable to perform pulmonary function tests: O2 saturation > 92% on room air (within 30 days prior to day 1 of protocol therapy)
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative), and syphilis rapid plasma reagin (RPR) (within 30 days prior to day 1 of protocol therapy)

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed OR
  * If seropositive for HIV, HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note: Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 30 days prior to day 1 of protocol therapy)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior allogeneic HCT
* Chemotherapy, radiation therapy, biological therapy, immunotherapy within 21 days prior to day 1 of protocol therapy

  * Note: Conditioning regimen within 21 days prior to day 1 of protocol therapy is not considered as an exclusion criterion. Patients on maintenance chemotherapy are not excluded
* Other investigational drugs for treatment of GVHD
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents
* Psychological issues, no appropriate caregivers identified, or non-compliant to medication
* Clinically significant uncontrolled illness
* Uncontrolled infection (bacterial, viral, fungal)
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Grade III-IV acute graft versus host disease (GVHD) | By day 100
  Acute GVHD will be graded and staged according to Mount Sinai Acute GVHD International Consortium (MAGIC) criteria.
GVHD-free relapse-free survival rate | From start of hematopoietic cell transplantation to grade III-IV acute GvHD, chronic GvHD requiring systemic treatment, relapse, or death (from any cause), whichever occurs first, assessed at 1 year
  Will be calculated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 2 years
  The toxicity/adverse event information recorded on each subject will include type, severity, duration, and attribution/ association with the study regimen. Tables will be constructed to summarize the observed incidence, severity and type of toxicity, including infection.
Overall survival | Day of stem cell infusion (day 0) until death or last follow-up, assessed at 100 days
  Will be calculated using the Kaplan-Meier method.
Overall survival | Day of stem cell infusion (day 0) until death or last follow-up, assessed at 180 days
  Will be calculated using the Kaplan-Meier method.
Overall survival | Day of stem cell infusion (day 0) until death or last follow-up, assessed at 1 year
  Will be calculated using the Kaplan-Meier method.
Progression free survival | From the date of stem cell infusion to the date of death, disease relapse/progression, or last follow-up, assessed at 100 days
  Will be calculated using the Kaplan-Meier method.
Progression free survival | From the date of stem cell infusion to the date of death, disease relapse/progression, or last follow-up, assessed at 180 days
  Will be calculated using the Kaplan-Meier method.
Progression free survival | From the date of stem cell infusion to the date of death, disease relapse/progression, or last follow-up, assessed at 1 year
  Will be calculated using the Kaplan-Meier method.
Relapse/progression | Day 0 to relapse/progression, assessed at 100 days
  The cumulative incidence will be calculated using the competing risk method.
Relapse/progression | Day 0 to relapse/progression, assessed at 180 days
  The cumulative incidence will be calculated using the competing risk method.
Relapse/progression | Day 0 to relapse/progression, assessed at 1 year
  The cumulative incidence will be calculated using the competing risk method.
Non-relapse mortality | Day 0 until non-disease related death or last follow-up, assessed at 100 days
  The cumulative incidence will be calculated using the competing risk method.
Non-relapse mortality | Day 0 until non-disease related death or last follow-up, assessed at 180 days
  The cumulative incidence will be calculated using the competing risk method.
Non-relapse mortality | Day 0 until non-disease related death or last follow-up, assessed at 1 year
  The cumulative incidence will be calculated using the competing risk method.
Rate of acute GVHD | On day 100
  Acute GVHD will be graded and staged according to MAGIC criteria. The first day of acute GVHD onset at a certain grade will be used to calculate the cumulative incidence (grades II-IV). The endpoint will be evaluated from day 0 through 100 days post-transplant. The cumulative incidence will be calculated using the competing risk method.
Rate of chronic GVHD | From day 80 through 1 year post-transplant
  Chronic graft versus host disease will be evaluated and scored according to National Institutes of Health Consensus Staging. The first day of chronic GVHD onset will be used to calculate the cumulative incidence. The cumulative incidence will be calculated using the competing risk method.
Rate of infection | Day -7 to day 120
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any. This data will be captured via case report form and will be collected from day -7 to day 120 post-transplant and will follow the same data collection intervals as the toxicity and adverse event data.
Rate of hematologic recovery | Up to 2 years
  Absolute neutrophil count >= 0.5 x 10^3/uL achieved and sustained for 3 consecutive lab values on different days with no subsequent decline.
  Platelets >= 20 K/uL independent of platelet transfusion support (date should reflect no transfusions in previous 7 days, and the first of 3 consecutive lab values on different days).
Incidence of cytokine release syndrome | Up to 2 years
  Defined and graded per American Society for Transplantation and Cellular Therapy criteria.
Gut microbiome assessment | Up to 2 years
  Gut microbiome diversity will be assessed by the inverse Simpson Index and compared among CBM588-treated/untreated patients; the inverse Simpson index is an ecological measure of α microbial diversity calculated by the inverse of the expected probability of 2 randomly selected bacterial sequences as belonging to the same operational taxonomic unit.

CONTACTS AND LOCATIONS:
Overall Officials: Monzr M Al Malki, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States